CLINICAL TRIAL: NCT02964676
Title: Clinical Efficacy and Safety of Minimally Invasive Glaucoma Surgery on Chinese Primary Angle Closure Glaucoma
Brief Title: Clinical Efficacy and Safety of Minimally Invasive Glaucoma Surgery on Primary Angle Closure Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YFZX2016002
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIT group (Experimental): PACG in AIT group will receive ab interno trabeculectomy with Trabectome and before AIT, Laser Peripheral Iridectomy (LPI) will be performed first.
  Interventions: Procedure: ab interno trabeculectomy with Trabectome
- Trab group (Active Comparator): PACG in AIT group will receive trabeculectomy.
  Interventions: Procedure: trabeculectomy

INTERVENTIONS:
Procedure: ab interno trabeculectomy with Trabectome — 123 PACG will be recruited to receive ab interno trabeculectomy with Trabectome and before this surgery, laser peripheral iridectomy will be performed firstly
  Arms: AIT group
Procedure: trabeculectomy — 123 PACG will be recruited to receive trabeculectomy to reduce IOP
  Arms: Trab group

SUMMARY:
To evaluate the clinical efficacy (intraocular pressure reduction , success rate, the number of antiglaucoma medication) and safety of ab interno trabeculectomy (AIT) with Trabectome in Chinese PACG .

DETAILED DESCRIPTION:
A randomized, single blind, positive parallel control study method was used.This prospective case series will recruit 246 Chinese POAG, 123 cases in the experimental group will receive AIT treatment and 123 cases in the control group will receive trabeculectomy(Trab) surgery.Measurements of intraocular pressure(IOP) , visual acuity, refraction, slit lamp examination of the anterior segment and fundus, optical coherence tomography(OCT) to detect retinal nerve fiber layer thickness, macular thickness, visual field, gonioscopy and ultrasonic biological microscopy (UBM) will be recorded.They will be followed up for 12 months. The main outcome is success rate of IOP reduction and the other outcome are the number of antiglaucoma medication and complications .

ELIGIBILITY:
Inclusion Criteria:

* Primary Angle Closure Glaucoma (PACG) with visible trabecular meshwork from 90︒ to 180︒ on gonioscopy and IOP couldn't be controlled ≤21mmHg with pilocarpine eye drop only.
* willing to accept the antiglaucoma surgery
* volunteer to participate in this study and be able to follow up on time
* previous antiglaucoma filtering surgery or laser surgery(LPI, SLT) and previous cataract surgery were not ruled out
* Exclusion Criteria:
* visual acuity lower than HM or central tubular visual field
* corneal edema or large pterygium affecting the observation of anterior angle
* the demarcation of the scleral process and trabecular meshwork is not clear on gonioscopy
* new vessels on the iris surface or in the anterior angle chamber
* the eye received surgery is the only eye with visual function, that is the contralateral eye is blind
* requiring long-term use of anticoagulant drugs for systemic reasons
* abnormal coagulation function
* with specific clear scar physique
* cannot participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
success rate of IOP reduction | 12 months
  IOP ≤21mmHg and IOP reduction rate ≥20% with or without antiglaucoma medications and without additional glaucoma surgery

SECONDARY OUTCOMES:
number of antiglaucoma medication | 12 months
  numbers of antiglaucoma medication will be recorded before surgery and 12 months follow up.
complication rate | 12 months
  all the complications related to the surgery will be evaluated and recorded.
24-hour IOP fluctuations | 12 months
  24-hour IOP fluctuations curve will be recorded before treatment and 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: LING GE, M.d., Principal Investigator — Shanghai Eye Disease Prevention and Treatment Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He M, Foster PJ, Ge J, Huang W, Zheng Y, Friedman DS, Lee PS, Khaw PT. Prevalence and clinical characteristics of glaucoma in adult Chinese: a population-based study in Liwan District, Guangzhou. Invest Ophthalmol Vis Sci. 2006 Jul;47(7):2782-8. doi: 10.1167/iovs.06-0051. PMID 16799014
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Palanca-Capistrano AM, Hall J, Cantor LB, Morgan L, Hoop J, WuDunn D. Long-term outcomes of intraoperative 5-fluorouracil versus intraoperative mitomycin C in primary trabeculectomy surgery. Ophthalmology. 2009 Feb;116(2):185-90. doi: 10.1016/j.ophtha.2008.08.009. Epub 2008 Oct 18. PMID 18930550
- [Background] Wang M, Fang M, Bai YJ, Zhang WZ, Lin MK, Liu BQ, Hao YT, Ling YL, Zhuo YH, Ge J. Comparison of combined phacotrabeculectomy with trabeculectomy only in the treatment of primary angle-closure glaucoma. Chin Med J (Engl). 2012 Apr;125(8):1429-33. PMID 22613648
- [Background] Wagn X, Jia C, Feng MY, Meng HL, Fan SJ, Xie LL, Sun LP, Liu LR, Xie C, Peng Y, Tang X, Liagn YB, Zhai G, Jiang YQ, Ye TC, Wang NL. [Assess correlation between bleb morphology at long-term intraocular pressure effect in primary angle-closure glaucoma following trabeculectomy]. Zhonghua Yan Ke Za Zhi. 2011 Oct;47(10):898-902. Chinese. PMID 22321499
- [Background] Wang M, Ge J, Lin MK, Zhuo YH, Ling YL, Fang M, Liu X, Peng SX, Yu MB. [Clinical observation of trabeculectomy for primary angle closure glaucoma]. Zhonghua Yan Ke Za Zhi. 2009 Apr;45(4):338-43. Chinese. PMID 19575967
- [Background] Sihota R, Gupta V, Agarwal HC. Long-term evaluation of trabeculectomy in primary open angle glaucoma and chronic primary angle closure glaucoma in an Asian population. Clin Exp Ophthalmol. 2004 Feb;32(1):23-8. doi: 10.1046/j.1442-9071.2004.00752.x. PMID 14746586
- [Background] Tsai HY, Liu CJ, Cheng CY. Combined trabeculectomy and cataract extraction versus trabeculectomy alone in primary angle-closure glaucoma. Br J Ophthalmol. 2009 Jul;93(7):943-8. doi: 10.1136/bjo.2008.151803. Epub 2009 Apr 20. PMID 19383599
- [Background] Wilson MR, Mendis U, Paliwal A, Haynatzka V. Long-term follow-up of primary glaucoma surgery with Ahmed glaucoma valve implant versus trabeculectomy. Am J Ophthalmol. 2003 Sep;136(3):464-70. doi: 10.1016/s0002-9394(03)00239-3. PMID 12967799
- [Background] Soltau JB, Rothman RF, Budenz DL, Greenfield DS, Feuer W, Liebmann JM, Ritch R. Risk factors for glaucoma filtering bleb infections. Arch Ophthalmol. 2000 Mar;118(3):338-42. doi: 10.1001/archopht.118.3.338. PMID 10721955
- [Background] DeBry PW, Perkins TW, Heatley G, Kaufman P, Brumback LC. Incidence of late-onset bleb-related complications following trabeculectomy with mitomycin. Arch Ophthalmol. 2002 Mar;120(3):297-300. doi: 10.1001/archopht.120.3.297. PMID 11879132
- [Background] Saheb H, Ahmed II. Micro-invasive glaucoma surgery: current perspectives and future directions. Curr Opin Ophthalmol. 2012 Mar;23(2):96-104. doi: 10.1097/ICU.0b013e32834ff1e7. PMID 22249233
- [Background] Ho CL, Lai JS, Aquino MV, Rojanapongpun P, Wong HT, Aquino MC, Gerber Y, Belkin M, Barkana Y. Selective laser trabeculoplasty for primary angle closure with persistently elevated intraocular pressure after iridotomy. J Glaucoma. 2009 Sep;18(7):563-6. doi: 10.1097/IJG.0b013e318193c2d1. PMID 19745672
- [Result] Mosaed S, Dustin L, Minckler DS. Comparative outcomes between newer and older surgeries for glaucoma. Trans Am Ophthalmol Soc. 2009 Dec;107:127-33. PMID 20126489
- [Result] Minckler D, Mosaed S, Dustin L, Ms BF; Trabectome Study Group. Trabectome (trabeculectomy-internal approach): additional experience and extended follow-up. Trans Am Ophthalmol Soc. 2008;106:149-59; discussion 159-60. PMID 19277230
- [Result] Vinod K, Gedde SJ. Ab interno trabeculectomy: patient selection and perspectives. Clin Ophthalmol. 2016 Aug 17;10:1557-64. doi: 10.2147/OPTH.S99746. eCollection 2016. PMID 27574396
- [Result] Minckler D, Baerveldt G, Ramirez MA, Mosaed S, Wilson R, Shaarawy T, Zack B, Dustin L, Francis B. Clinical results with the Trabectome, a novel surgical device for treatment of open-angle glaucoma. Trans Am Ophthalmol Soc. 2006;104:40-50. PMID 17471324
- [Result] Maeda M, Watanabe M, Ichikawa K. Evaluation of trabectome in open-angle glaucoma. J Glaucoma. 2013 Mar;22(3):205-8. doi: 10.1097/IJG.0b013e3182311b92. PMID 23429629
- [Result] Werth JP, Gesser C, Klemm M. [Diverse effectiveness of the trabectome for different types of glaucoma]. Klin Monbl Augenheilkd. 2015 Jan;232(1):72-8. doi: 10.1055/s-0034-1383010. Epub 2014 Oct 1. German. PMID 25272084
- [Result] Lee JWY, Yick DWF, Tsang S, Yuen CYF, Lai JSM. Efficacy and Safety of Trabectome Surgery in Chinese Open-Angle Glaucoma. Medicine (Baltimore). 2016 Apr;95(15):e3212. doi: 10.1097/MD.0000000000003212. PMID 27082559
- [Result] Jea SY, Mosaed S, Vold SD, Rhee DJ. Effect of a failed trabectome on subsequent trabeculectomy. J Glaucoma. 2012 Feb;21(2):71-5. doi: 10.1097/IJG.0b013e31820bcfda. PMID 21336149
- [Result] Huang P, Wang H, Wu H, Sun Y, Wang M, Cui Y, Qiu W, Yang Y, Ren Z, Zhang C, Wang N. [Preliminary investigation on the safety and efficacy of Trabectome]. Zhonghua Yan Ke Za Zhi. 2015 Feb;51(2):115-9. Chinese. PMID 25908002
- [Result] Bussel II, Kaplowitz K, Schuman JS, Loewen NA; Trabectome Study Group. Outcomes of ab interno trabeculectomy with the trabectome by degree of angle opening. Br J Ophthalmol. 2015 Jul;99(7):914-9. doi: 10.1136/bjophthalmol-2014-305577. Epub 2014 Oct 21. PMID 25336577